CLINICAL TRIAL: NCT06566820
Title: A Phase 3 Open Label Continuation Protocol of a Fixed Dose Combination of Aroxybutynin and Atomoxetine (AD109) in Obstructive Sleep Apnea
Brief Title: Continuation Protocol for Obstructive Sleep Apnea (OSA)
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APC-APN-306
Record Dates: First submitted 2024-07-03; First posted 2024-08-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: OSA
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AD109 (Experimental): Open Label AD109
  Interventions: Drug: Aroxybutynin and Atomoxetine

INTERVENTIONS:
Drug: Aroxybutynin and Atomoxetine — Fixed Dose Combination
  Other Names: AD109

SUMMARY:
The combination drug composed of aroxybutynin and atomoxetine, designated AD109, is being developed by Apnimed for the treatment of obstructive sleep apnea (OSA). The present study is a Phase 3 open label continuation protocol enrolling qualifying participants who completed one of the parent Phase 3 double-blind placebo-controlled studies, APC-APN-304 or APC-APN-305.

ELIGIBILITY:
Inclusion Criteria:

* Completion of APC-APN-304 without permanent discontinuation of IMP.
* Completion of APC-APN-305 without permanent discontinuation of IMP.

Exclusion Criteria:

* Participants are excluded from the study if participation would be considered unsafe by the investigator based on the individual's current status.
* Participants are excluded from the study if participation would be considered unsafe by the investigator based on concomitant therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1280 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AES) and Serious Adverse Events (SAEs) | through study completion, an average of 1 year
  An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. An SAE was an AE during any study phase that fulfills one or more of the following criteria: results in death, life threatening (The term 'life-threatening' in the definition of 'serious' refers to an event in which the participant was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe), requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity.
Number of Participants With Vital Signs Abnormalities | through study completion, an average of 1 year
  Vital signs that are planned to be assessed include parameters such as weight,heart rate and systolic and diastolic blood pressure.
Number of Participants With Concomitant Therapy (Medication or Devices) | through study completion, an average of 1 year
  Concomitant therapy with devices (i.e., CPAP) and concomitant medications are other prescription medications, over-the-counter (OTC) drugs or dietary supplements that a study participant takes in addition to the drug under investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Farkas, MD, Study Director — Apnimed
Locations (99):
- United States (93):
  - Sleep Disorders Center of America, Birmingham, Alabama
  - The University of Alabama/Institute for Rural Health Research, Tuscaloosa, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - Desert Clinical Reserach, LLC/CCT Research, Mesa, Arizona
  - Foothills Research Center/CCT Research, Phoenix, Arizona
  - Fiel Family and Sports Medicine/CCT Research, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Orange County Research Institute, Anaheim, California
  - Core Healthcare Group, Cerritos, California
  - Exalt Clinical Research, Inc., Chula Vista, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Santa Monica Clinical Trials, Los Angeles, California
  - Empire Clinical Research, Pomona, California
  - Probe Clinical Research Corporation, Riverside, California
  - Pacific Research Network, San Diego, California
  - TriValley Sleep Center, San Ramon, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Providere Research Inc., West Covina, California
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - Meris Clinical Research, Brandon, Florida
  - Teradan Clinical Trials, Brandon, Florida
  - St. Francis Medical Institute, Clearwater, Florida
  - Nouvelle Clinical Research, Cutler Bay, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Canvas Clinical Research, Lake Worth, Florida
  - Florida Lung & Sleep Associates, Lehigh Acres, Florida
  - Ivetmar Medical Group, LLC, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - PharmaDev Clinical Research Institute, LLC, Miami, Florida
  - Flourish Research, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - JSV Clinical Research Study Inc., Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Central Florida Pediatric Sleep Disorders d/b/a Florida Pediatric Institute, LLC, Winter Park, Florida
  - Clinical Site Partners, LLC dba Flourish Research, Winter Park, Florida
  - Neurotrials Research Inc, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Georgia Neurology and Sleep Medicine Associates, Suwanee, Georgia
  - Medster Research, Valdosta, Georgia
  - St. Luke's Idaho Pulmonary Associates - Meridian Clinic, Meridian, Idaho
  - Chicago Research Center, Inc., Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Advanced ENT and Allergy, Louisville, Kentucky
  - Centennial Medical Group Research Department, Columbia, Maryland
  - Sleep Disorders Centers of the Mid-Atlantic, Glen Burnie, Maryland
  - Velocity Clinical Research, Rockville, Maryland
  - Neurocare, Inc., Newton, Massachusetts
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - Baystate Clinical Trials Unit, Springfield, Massachusetts
  - University of Michigan Clinical Research Unit, Ann Arbor, Michigan
  - Revive Research Institute, Inc., Lathrup Village, Michigan
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - Clinical Neurophysiology Services PC, Sterling Heights, Michigan
  - Sleep Medicine and Research Center, St. Luke's Hospital, Chesterfield, Missouri
  - Healthcare Research Network, Hazelwood, Missouri
  - Clayton Sleep Institute, LLC, St Louis, Missouri
  - Henderson Clinical Trials, Henderson, Nevada
  - Las Vegas Clinical Trials, LLC, North Las Vegas, Nevada
  - Clinilabs Drug Development Corporation, Eatontown, New Jersey
  - Sleep Dynamics, Neptune City, New Jersey
  - Maimonides Sleep Arts & Sciences, Albuquerque, New Mexico
  - Northwell Health, New Hyde Park, New York
  - Research Carolina Elite, Denver, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Peters Medical Research LLC, High Point, North Carolina
  - Advanced Respiratory and Sleep Medicine, Huntersville, North Carolina
  - Coastal Carolina Health Care, P.A. Pulmonary and Sleep Medicine, New Bern, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - NeuroScience Research Center, LLC, Canton, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Intrepid Research, LLC, Cincinnati, Ohio
  - Northwest Research Center, Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - Respiratory Specialists, Wyomissing, Pennsylvania
  - Lowcountry Lung and Critical Care, PA, Charleston, South Carolina
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Velocity Clinical Research, Greenville, Greenville, South Carolina
  - OnSite Clinical Solutions, LLC, Rock Hill, South Carolina
  - Chattanooga Research & Medicine, Chattanooga, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Memorial Hermann Village, Houston, Texas
  - Houston Clinical Research Associates, Houston, Texas
  - Huntsville Research Institute, Huntsville, Texas
  - Sleep Therapy and Research Center, San Antonio, Texas
  - Element Research Group, San Antonio, Texas
  - South Ogden Family Medicine/CCT Research, South Ogden, Utah
  - Sleep Disorder Center of the Mid-Atlantic, Vienna, Virginia
- Canada (6):
  - Medical Arts Health Research Group, Kelowna, British Columbia
  - AMNDX Inc, Markham, Ontario
  - West Ottawa Sleep Centre, Ottawa, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Jodha Tishon, Inc., Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No